CLINICAL TRIAL: NCT03729115
Title: Chicago Alternative Prevention Study for Diverse Populations of High Risk Women
Brief Title: A Multi-Modality Surveillance Program for Women at High Risk for Breast Cancer
Acronym: CAPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB18-0970
Record Dates: First submitted 2018-10-12; First posted 2018-11-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening Arm (Other): Enrolled patients will undergo Magnetic Resonance Imaging (MRI) every 6 months (2x/year) in addition to an annual screening mammogram.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — Patients will have MRI scans every 6 months.

SUMMARY:
This study is aimed to establish a registry of women undergoing intensive surveillance for the early detection of breast cancer in high-risk women.

ELIGIBILITY:
Inclusion Criteria:

- Known BRCA1 or BRCA2, TP53, PALB2, PTEN, CDH1 and STK11 carrier. Women with pathogenic mutations in any other cancer susceptibility genes are eligible only if they also have a high PRS.

OR

* With life time risk of 30% or higher, based on Polygenic Risk Score that integrates genetic and non-genetic factors OR
* 5-years risk ≥ 6% for women 40-64 OR
* 5-years risk ≥ 6% for women 65+ AND breast density C or D AND a lifetime risk >= 20% (BCSC+PRS LTR or Tyrer-Cuzick LTR) OR
* Patients with history of chest wall radiation received before age 35. OR
* To promote health equity, women of African Ancestry < 45 years with at least one 1st or 2nd degree relative with breast or ovarian cancer are eligible because PRS Scores are not currently reported for AA women.
* Must be at least 25 years old.
* Willing to travel to participating site for imaging studies as well as any necessary follow-up procedures.
* Be able to give informed consent.

  * Patients with prior history of breast or ovarian cancer are eligible if they have completed all active treatments and are cancer free for two years.

Exclusion Criteria

* Undergoing active cancer treatment at the time of enrollment.
* Current pregnancy or plans for pregnancy within two years of enrollment.
* Presence of a pacemaker or any other metallic foreign object in their body that interferes with an MRI.
* Breast surgery within two weeks of study entry.
* Women with history of bilateral mastectomy are not eligible
* History of kidney disease or abnormal kidney function.
* History of dye allergy unless it can be mediated with antihistamines and/or steroids

  * Women can be taking hormone replacement therapy, tamoxifen, raloxifene, aromatase inhibitors, Parp Inhibitors as adjuvant therapy or participating in a chemoprevention trial.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of faster MRI protocols for a for a Personalized Risk-based Imaging Surveillance Model for diverse populations of high risk women. | 5 years
  We will test whether an abbreviated MRI (AB-MRI) is diagnostically equivalent to a full MRI. Eligible women will be scanned every 6 months with a full protocol MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Olufunmilayo I Olopade, MD, Principal Investigator — University of Chicago
Locations (1):
- University Of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States